CLINICAL TRIAL: NCT06627530
Title: A Randomized Trial of Neoadjuvant Leuprorelin, Darolutamide or Both Prior to Radical Prostatectomy for Intermediate or High-risk Prostate Cancer
Brief Title: COACTION Trial - COmbination Androgen bloCkade in inTermediate to hIgh-risk prOstate caNcer
Acronym: COAction
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brazilian Clinical Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001/2024
Record Dates: First submitted 2024-09-12; First posted 2024-10-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy; Darolutamide; Neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Leuprolide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Darolutamide + ADT leuprorelin (Experimental)
  Interventions: Drug: Darolutamide Oral Tablet; Drug: leuprorelin
- Darolutamide (Active Comparator)
  Interventions: Drug: Darolutamide Oral Tablet
- Leuprorelin (Active Comparator)
  Interventions: Drug: leuprorelin

INTERVENTIONS:
Drug: Darolutamide Oral Tablet — darolutamide 600 mg PO BID for 24 weeks
  Arms: Darolutamide; Darolutamide + ADT leuprorelin
Drug: leuprorelin — leuprorelin depot 22.5 mg SC every 12 weeks
  Arms: Darolutamide + ADT leuprorelin; Leuprorelin

SUMMARY:
A Randomized Trial of Neoadjuvant Leuprorelin, Darolutamide or Both Prior to Radical Prostatectomy for Intermediate or High-risk Prostate Cancer. Prospective, randomized, parallel group, open-label with blinded endpoint adjudication multicenter clinical trial.To assess, among patients with unfavorable intermediate to high-risk prostate cancer, whether a neoadjuvant combined treatment with leuprorelin (Leuprorelin) and darolutamide is superior to monotherapy in terms of complete or almost complete pathological response.A total of 144 patients with unfavorable intermediate to high-risk prostate cancer scheduled for radical prostatectomy with extended pelvic lymph node dissection will be randomized 1:1:1 to oral darolutamide, SC leuprorelin (Leuprorelin) or both (48 patients per arm) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years of age;
* Histologically confirmed unfavorable intermediate or high/very high risk non metastatic (by conventional imaging) prostate adenocarcinoma intended for surgery without neuroendocrine differentiation or small cell features;
* Unfavorable intermediate-risk:

  * ISUP grade 3, and/or > 50% positive biopsy cores and/or at least two intermediate-risk factors. Intermediate-risk factors:

    * Clinical tumor stage T2b or T2c (MRI based);
    * ISUP grade 2 or 3;
    * Prostate-specific antigen (PSA) level of 10-20 ng/mL.
* High-risk or very high-risk:

  * ≥cT3a (MRI based) or ISUP 4-5 or PSA>20 ng/mL;
  * cN1.
* ECOG 0-1;
* Baseline testosterone > 230 ng/dL;
* No prior prostate cancer treatment;
* Sexually active male subjects must agree to use condoms as an effective barrier method and refrain from sperm donation, and/or their female partners of reproductive potential to use a method of effective birth control, during the treatment with darolutamide and for 1 week after the end of treatment with darolutamide to prevent pregnancy;
* Written informed consent.

Exclusion Criteria:

* Unresectable prostate cancer;
* Histology of small cell carcinoma prostate cancer or adenocarcinoma with neuroendocrine features;
* Any prior prostate cancer treatment;
* Any active infection requiring IV antibiotics;
* Known additional malignancy that has a life-expectancy < 2 years;
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, heart failure with New York Heart Association Class Functional III or IV;
* Uncontrolled severe hypertension as indicated by a resting systolic BP ≥ 180 mmHg or diastolic BP ≥ 110 mmHg despite medical management;
* A gastrointestinal (GI) disorder or procedure which is expected to interfere significantly with absorption of darolutamide;
* Inability to swallow oral medications;
* Receipt of medications (e.g. finasteride, dutasteride) or agents that are likely to alter serum PSA levels within <= 42 days or 5 half-lives prior to registration, whichever is shorter.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with minimal residual disease | Patients are expected to undergo surgery after no more than 30 days after completion of the neoadjuvant regimen therapy, which will last for 24 weeks after randomization in all 3 groups.
  Proportion of patients with minimal residual disease, defined as residual cancer burden (RCB) ≤ 0.25 cm3 (tumor volume ≤ 0.5 cm3 × tumor cellularity ≤ 50%) or complete pathological response, assessed by pathology of surgical specimen obtained from prostatectomy.

SECONDARY OUTCOMES:
Complete biochemical response assessed by serum PSA with the rate of PSA<0,2 ng/dL | 24 weeks
Treatment emergent adverse events and serious adverse events. | 24 weeks
PSA levels at 3 months after prostatectomy. | in 42 weeks
Testosterone levels. | in 42 weeks
Number of positive lymph nodes. | 30 weeks
Number of positive surgical margins. | 30 weeks
Perioperative complications. | 42 weeks
Quality of life using IEEF5 and HRQoL questionnaires pre and post neoadjuvant treatment. | 42 weeks
Downstaging (changes in TNM - Classification of Malignant Tumours stage) based on surgical specimen. | 30 weeks
  Prostate cancer TNM (Classification of Malignant Tumours) staging AJCC (American Joint Committee on Cancer) UICC (Union for International Cancer Control) 8th edition

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C Maluf, MD, Study Chair — Brazilian Clinical Research Institute
Locations (6):
- Brazil (6):
  - Santa Casa de Misericórdia de Feira de Santana, Feira de Santana, Estado de Bahia
  - Hospital Ophir Loyola, Belém, Pará
  - Hospital São Marcos, Teresina, Piauí
  - Hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clínicas Ijuí, Ijuí, Rio Grande do Sul
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo, São Paulo